CLINICAL TRIAL: NCT03869593
Title: Role of the NLRP3 Inflammasome in Escherichia Coli and Staphylococcus Aureus Bacteria
Acronym: NLRP3-Bact
Status: Terminated | Type: Observational
Why Stopped: End of recruitment period
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 18-AOI-08
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Escherichia Coli Infections; Staphylococcus Aureus
MeSH Terms: conditions — Escherichia coli Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 samples of blood will be collected during a routine blood test. A sample will allow the analysis of the study, the second will join a biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting E. coli and S. aureus bacteremia: Here, to determine the importance of the mutation we will analyze the blood content of patients presenting E. coli and S. aureus bacteremia
  Interventions: Genetic: Sample analysis

INTERVENTIONS:
Genetic: Sample analysis — Here, to determine the importance of the mutation we will analyze the blood content of patients presenting E. coli and S. aureus bacteremia

SUMMARY:
Our previous studies delineate a novel pathway of immune activation in animals that the investigators have named Anti-Virulence Immunity (AVI). Using a mice model of bacteremia, the investigators have demonstrated that Escherichia coli Cytotoxic Necrotizing Factor 1 (CNF1) activity is sensed by the immune system. This immune sensing results in a rapid bacterial clearing during bacteremia triggered by uropathogenic E. coli-expressing CNF1. The investigators already confirmed the involvement of one inflammasome using macrophages isolated from Knock-out mice. The investigators have recently determined the conservation in human monocytes of the interleukin -1beta maturation triggered by CNF1 and observed the heterogeneous capacity of monocytes to respond to the CNF1 treatment depending on the donors. Here, to determine the importance in natura of AVI the investigators will analyze the blood content of patients presenting E. coli and S. aureus bacteremia. The DNA of monocytes isolated from patients will be extracted and various genes implicated in the activity of various inflammasomes will be sequenced to identify mutations that could explain the susceptibility to bacteremia or a specific clinical presentation, i.e. requirement of a management in ICU because of organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with S. aureus or E. coli bacteriostatic bacteremia defined by at least one positive blood culture bottle
* Patient requiring a blood test as part of his bacteremia
* not subject to a judicial protection measure
* Signature of the non-opposition of consent (for minor patients signed by one of the parents or the representative of the parental authority)
* Affiliation to social security

Exclusion Criteria:

* Immunocompromised patient defined by:

  * current immunosuppressive therapies: corticosteroids, chemotherapy, biotherapy
  * solid organ transplant patient or hematopoietic stem cell transplant
  * chemotherapy-induced neutropenia
  * Congenital immune deficiency
* bacteremia related to a peripheral or central catheter
* Urinary obstruction not lifted within the first 24 hours of management
* Intra-abdominal infection collected undrained in the first 24 hours of management
* primary infectious focus represented by mechanically ventilated pneumonia
* Pregnant or lactating woman

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with S. aureus or E. coli bacteremia defined by at least one positive blood culture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Establish an association between mutations in some inflammasomes and occurrence of E. coli associated with sepsis. | 1 hour
Establish an association between mutations in some inflammasomes and occurrence of S. aureus bacteremia associated with sepsis. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Johan COURJON, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (3):
- France (3):
  - CHG d'Antibes, Antibes
  - CH Pierre Nouveau, Cannes
  - CHU de Lenval, Nice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CC, Chen SY, Chang IJ, Chen SC, Wu SC. Comparison of clinical manifestations and outcome of community-acquired bloodstream infections among the oldest old, elderly, and adult patients. Medicine (Baltimore). 2007 May;86(3):138-44. doi: 10.1097/SHK.0b013e318067da56. PMID 17505253
- [Background] Weinstein MP, Towns ML, Quartey SM, Mirrett S, Reimer LG, Parmigiani G, Reller LB. The clinical significance of positive blood cultures in the 1990s: a prospective comprehensive evaluation of the microbiology, epidemiology, and outcome of bacteremia and fungemia in adults. Clin Infect Dis. 1997 Apr;24(4):584-602. doi: 10.1093/clind/24.4.584. PMID 9145732
- [Background] Wisplinghoff H, Bischoff T, Tallent SM, Seifert H, Wenzel RP, Edmond MB. Nosocomial bloodstream infections in US hospitals: analysis of 24,179 cases from a prospective nationwide surveillance study. Clin Infect Dis. 2004 Aug 1;39(3):309-17. doi: 10.1086/421946. Epub 2004 Jul 15. PMID 15306996
- [Background] Valles J, Palomar M, Alvarez-Lerma F, Rello J, Blanco A, Garnacho-Montero J, Martin-Loeches I; GTEI/SEMICYUC Working Group on Bacteremia. Evolution over a 15-year period of clinical characteristics and outcomes of critically ill patients with community-acquired bacteremia. Crit Care Med. 2013 Jan;41(1):76-83. doi: 10.1097/CCM.0b013e3182676698. PMID 23222266
- [Background] Herrmann JB, Muenstermann M, Strobel L, Schubert-Unkmeir A, Woodruff TM, Gray-Owen SD, Klos A, Johswich KO. Complement C5a Receptor 1 Exacerbates the Pathophysiology of N. meningitidis Sepsis and Is a Potential Target for Disease Treatment. mBio. 2018 Jan 23;9(1):e01755-17. doi: 10.1128/mBio.01755-17. PMID 29362231